CLINICAL TRIAL: NCT04856449
Title: A Pilot Randomized-controlled Study of Dialectical Behavioral Skills Training Plus EMDR for Borderline Personality Disorder and Trauma
Brief Title: DBT Skills Plus EMDR for BPD and Trauma
Acronym: TT-BPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: EMDR Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIBSP-TLP-2020-105
Record Dates: First submitted 2021-04-08; First posted 2021-04-23 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Borderline Personality Disorder; Trauma
MeSH Terms: conditions — Borderline Personality Disorder; Wounds and Injuries | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT Skills Training (Experimental): This intervention will consist of a 6-month-group DBT-skills training continuation, in which participants will be trained in mindfulness, emotion regulation, distress tolerance and interpersonal effectiveness.
  Interventions: Behavioral: Dialectical Behavioral Therapy Skills Training
- Eye Movement Desensitization and Reprocessing (EMDR) (Active Comparator): EMDR will consist of individual therapy sessions that will be focused on processing traumatic memories. Participants will receive up to 16 individual EMDR sessions, of 60 min each.
  Interventions: Behavioral: EMDR

INTERVENTIONS:
Behavioral: Dialectical Behavioral Therapy Skills Training — DBT skills training consists of a 6 months training in mindfulness, emotion regulation, interpersonal effectiveness and distress tolerance.
  Other Names: DBT-ST
  Arms: DBT Skills Training
Behavioral: EMDR — EMDR sessions will be conducted to reprocess trauma-related memories.
  Arms: Eye Movement Desensitization and Reprocessing (EMDR)

SUMMARY:
Borderline Personality Disorder (BPD) is a severe disorder that frequently co-occurs with post-traumatic stress disorder (PTSD). The comorbidity of BPD and PTSD is more disabling, predicting lower rates of BPD remission. Dialectical behavioral skills training (DBT-ST), is a group-delivered training that covers four types of skills: emotion regulation, mindfulness, interpersonal effectiveness and distress tolerance. As a stand-alone treatment, research suggest that DBT-ST is an efficacious treatment for BPD. In parallel, EMDR has emerged in last years as an efficacious approach to adult trauma. However, so far, the efficacy of EMDR to treat trauma in populations with BPD diagnosis has not been tested. The present pilot randomized-controlled clinical trial aims to test whether a combination of DBT-ST plus EMDR could be efficacious to treat trauma in individuals with BPD. 40 participants will be recruited from the BPD Unit at the Hospital de la Santa Creu I Sant Pau (Barcelona, Spain) and will be randomized (1:1) to DBT-ST + EMDR or DBT-ST alone. The primary outcome will be the reduction of PTSD symptoms. In addition, symptom-related variables will be collected before and after the interventions. This will be the first study to test the combination of DBT-ST and EMDR.

ELIGIBILITY:
Inclusion Criteria:

* men and women between 18 and 60 years old
* having had adverse childhood experiences and/or current PTSD symptoms
* signed informed consent

Exclusion Criteria:

* lifetime diagnosis of schizophrenia, drug-induced psychosis, organic brain syndrome, bipolar disorder, or mental retardation.
* participation in any psychotherapy during the study or having received DBT or EMDR in the past

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Borderline Symptom List 23 (BSL-23) | 1 week
  The scores range from a 0 to 4, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Impact of Events Scale Revised | 1 week
  The scores range from a 0 to 25, with higher scores indicating a higher impact of the traumatic event (worse outcome)
Patient Health Questionnaire (PHQ-9) | 2 weeks
  The scores range from a 0 to 27, with higher scores indicating a worse outcome.
DISSOCIATIVE EXPERIENCES SCALE (DES) | 1 month
  The scores range from 0 to 100, with higher scores representing a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No